CLINICAL TRIAL: NCT02357992
Title: STARS Revised Clinical Trial Protocol: Stereotactic Ablative Radiotherapy (SABR) in Stage I Non-small Cell Lung Cancer Patients Who Can Undergo Lobectomy
Brief Title: Lung Cancer STARS Trial - STARS Revised Clinical Trial Protocol: Stereotactic Ablative Radiotherapy (SABR) in Stage I Non-small Cell Lung Cancer Patients Who Can Undergo Lobectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Varian Medical Systems (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007-0870; NCI-2015-00536 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2015-02-03; First posted 2015-02-06 (Estimated); Results first posted 2022-10-14 (Actual); Last update posted 2022-10-14 (Actual); Status verified 2022-10

CONDITIONS: Lung Cancer
Keywords: Lung cancer; Non-small cell lung cancer; NSCLC; Squamous cell carcinoma; Adenocarcinoma with or without BAC features; Large cell carcinoma with or without neuroendocrine features; Neuroendocrine carcinoma; Bronchioloalveolar cell carcinoma; Stereotactic radiotherapy (SRT); SRT; Stereotactic ablative radiotherapy; SABR; Radiation therapy; XRT
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Carcinoma, Squamous Cell; Carcinoma, Neuroendocrine | interventions — Radiosurgery; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Stereotactic Radiotherapy (SRT) (Experimental): Participants receive stereotactic body radiotherapy (SABR) once a day for 3-4 days in a row.
  50Gy delivered in 4 fractions for central tumor, or 54Gy delivered in 3 fractions for peripheral tumor.
  Interventions: Radiation: Stereotactic Body Radiotherapy (SABR)

INTERVENTIONS:
Radiation: Stereotactic Body Radiotherapy (SABR) — SABR once a day for 3-4 days in a row, 50Gy in 4 fractions for central tumor, or 54Gy in 3 fractions for peripheral tumor.
  Other Names: SABR; XRT; Radiation therapy

SUMMARY:
The goal of this clinical research study is to evaluate the outcome of a standard radiation treatment called stereotactic radiotherapy (SRT) for NSCLC.

Specifically, researchers want to learn if standard SRT has as good of an outcome at 3 years after the procedure. The safety of the study treatment will also be analyzed.

DETAILED DESCRIPTION:
The Study Treatment:

The treatment being used in this study is considered standard, but researchers want to see its outcome in early-stage NSCLC.

The radiation (SRT) in this study is designed to kill tumor cells by using beams of radiation aimed directly at the tumor from different angles. The doctor uses computed tomography (CT) scans to plan exactly where to direct the beams to go. A computer is used to show the location, size, and shape of the tumor. SRT is designed to cause less damage to normal tissue than surgery, and it also may allow a higher dose of radiation to be given to the tumor than if other forms of radiation therapy were used.

The SRT in this study will be performed using a radiation machine called Linear Accelerator (Linac).

Study Group:

If you are found to be eligible to take part in this study, you will receive SRT (as an out-patient) once a day for 3-4 days in a row. You will be asked to hold still during the entire treatment (for about 1 to 1 1/2 hours each time). The machine will move around you, but you will not see or feel anything (similar to getting an x-ray).

Follow-Up Visits:

During the treatment period, you will be seen by a doctor and/or research nurse in order to check for any side effects. A physical exam will be performed, and your medical history will be recorded. These follow-up procedures will be done once on any day of your SRT.

A physical exam will be performed and your medical history will be recorded at 6 and 12 months, then at 1 1/2, 2, 3, 4, and 5 years after your SRT. If the doctor decides it is necessary, you will have a chest x-ray to check the status of the disease.

At 6 to 12 months after SRT, you will have either a PET-CT scan or CT scan to check the status of the disease.

At 1 year after SRT, you will have breathing tests to check your lung function. You will also have a CT scan to check the status of your disease.

At 1 1/2 year and then at 2, 3, 4, and 5 years after SRT, you will have a CT scan to check the status of your disease.

Possible Re-Treatment On Study:

If one of your follow-up CT scans shows that the tumor has come back in the same location or very close, you will have a PET scan and a tumor biopsy. The purpose is to confirm the status of the disease. To collect a tumor biopsy, the affected area is numbed with anesthetic, and a small amount of tissue is withdrawn through a large needle.

As soon as the results of the scan and biopsy come back, the study doctor will discuss with you the different treatment options. You may receive surgery, radiation therapy, or chemotherapy, depending on the status of the disease. You will receive a separate consent form that describes the treatment in more detail, as well as the risks.

After this "re-treatment", you will stay on the same schedule for study follow-up visits as you were following before.

Length of Study Participation:

Your participation in this study will be over after the 5-year follow-up visit.

This is an investigational study. The treatment is commercially available and considered standard for early-stage NSCLC. This includes the use of the Linac radiation machine, which is FDA approved and commercially available.

Up to 80 treated patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Histological confirmation of non-small cell cancer will be required by either biopsy or cytology. The following primary cancer types are eligible: squamous cell carcinoma, adenocarcinoma with or without BAC features, large cell carcinoma with or without neuroendocrine features, neuroendocrine carcinoma, bronchioloalveolar cell carcinoma, or non-small cell carcinoma not otherwise specified.
2. Eligible patients must have appropriate staging studies identifying them as specific subsets of the revised IASLC stage IA based on the following combination of TNM staging: T1a,N0,M0 or T1b,N0,M0
3. A PET/CT scan is required. Patients with hilar or mediastinal lymph nodes with short axis diameter </= 1cm and no abnormal hilar or mediastinal uptake on PET will be considered N0. Patients with > 1 cm short axis diameter of hilar or mediastinal lymph nodes on CT or abnormal PET (including suspicious but non-diagnostic uptake) may still be eligible if directed tissue biopsy of all abnormally identified areas are negative for cancer. Solitary pulmonary lesions </= 6mm will not be considered significant.
4. Patients must be considered a candidate for surgical resection of the primary tumor. Standard justification for deeming a patient medically operable based on pulmonary function for surgical resection of NSCLC may include any of the following: Baseline FEV1 > 40% predicted, post-operative predicted FEV1 > 30% predicted, diffusion capacity > 40% predicted, absent baseline hypoxemia and/or hypercapnia, exercise oxygen consumption > 50% predicted, absent severe pulmonary hypertension, absent severe cerebral, cardiac, or peripheral vascular disease, and absent severe chronic heart disease.
5. Patients must be >/= 18 years of age.
6. The patient's Zubrod performance status must be Zubrod 0-2.
7. PET/CT scan to include both lungs, the mediastinum, and adrenal glands; Primary tumor dimension will be measured on diagnostic CT and again on simulation CT. Must be done within 10 weeks prior to study entry.
8. Mediastinoscopy or endobronchial ultrasound (EBUS) guided biopsy of mediastinal lymph nodes is required for all patients. Must be done within 10 weeks of study entry.
9. MRI or CT scans of Brain if there are symptoms or signs suggesting brain metastases, must be done within 10 weeks prior to study entry.
10. Invasive Mediastinal Staging - All patients with CT and/or PET evidence of hilar (level 10) or mediastinal lymph nodes > 1.0 cm in the shortest diameter must be staged by either cervical mediastinoscopy, esophageal endoscopic ultrasound guided biopsy, or endobronchial ultrasound guided biopsy.
11. Patients must sign a study-specific consent form.
12. Patients (men and women) of child bearing potential should use an effective (for them) method of birth control throughout their participation in this study.

Exclusion Criteria:

1. Patients with primary tumors > 3 cm.
2. Patients with well-differentiated neuroendocrine carcinoma (carcinoid tumor).
3. Direct evidence of regional or distant metastases after appropriate staging studies, or synchronous primary or prior malignancy in the past 3 years other than nonmelanomatous skin cancer or in situ cancer.
4. Previous lung or mediastinal radiotherapy.
5. Plans for the patient to receive other concomitant local therapy (including standard fractionated radiotherapy and surgery) while on this protocol except at disease progression.
6. Pregnant or lactating women, as treatment involves unforeseeable risks to the embryo or fetus.
7. Cannot achieve acceptable SABR planning to meet minimal requirement of target coverage and dose-volume constraints of critical structures (see RT techniques).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2010-04-05 (Actual); Primary Completion 2021-09-17 (Actual); Study Completion 2021-09-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jack Roth, MD, BA, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Chang JY, Mehran RJ, Feng L, Verma V, Liao Z, Welsh JW, Lin SH, O'Reilly MS, Jeter MD, Balter PA, McRae SE, Berry D, Heymach JV, Roth JA; STARS Lung Cancer Trials Group. Stereotactic ablative radiotherapy for operable stage I non-small-cell lung cancer (revised STARS): long-term results of a single-arm, prospective trial with prespecified comparison to surgery. Lancet Oncol. 2021 Oct;22(10):1448-1457. doi: 10.1016/S1470-2045(21)00401-0. Epub 2021 Sep 13. PMID 34529930
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: April 2010- January 2018.
Pre-assignment Details: A total of 122 participants were consented; 6 were screen failures.
Groups:
- Surgery (S) vs. SBRT: These patients were randomized to surgery vs. SBRT. Both open thoracotomy and video assisted thoracotomy (VATS) are acceptable procedures. Surgery may consist of a lobectomy, sleeve resection, bilobectomy or pneumonectomy as determined by the attending surgeon based on the operative findings. The type of resection chosen should provide complete removal of the primary lesion with negative gross and microscopic margins. Documentation of margins (bronchial and vascular and any other required) by frozen sections at surgery is recommended. Limited resection including wedge or segmental resections should not be performed unless there are unforeseen problems at the time of surgery.
- Stereotactic Body Radiation Therapy (SBRT) (R): SBRT for lung cancer utilizes elements of 3-DCRT and also incorporates a variety of systems for taking cancer motion into consideration and decreasing set-up uncertainty using image guided radiotherapy techniques (9). These systems allow reduction of treatment volumes facilitating hypofractionation with markedly increased daily doses (>10 GY) and a significantly reduced overall treatment time. The combination of multiple beam angles to achieve sharp dose gradients, high precision localization and a high dose per fraction in extracranial locations are referred to as SBRT. This approach delivers a high biological effective dose (BED) to the target while minimizing the normal tissue toxicities, this may translate into improved local control and survival.
Period: Overall Study
Arm/Group | Surgery (S) vs. SBRT | Stereotactic Body Radiation Therapy (SBRT) (R)
Started | 36 | 80
Completed | 36 | 80
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Surgery (S) vs. SBRT | Stereotactic Body Radiation Therapy (SBRT) (R) | Total
Number analyzed (Participants) | 36 | 80 | 116
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 22 | 38
  >=65 years | 20 | 58 | 78
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 36 | 54
  Male | 18 | 44 | 62
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 5 | 5
  Not Hispanic or Latino | 14 | 70 | 84
  Unknown or Not Reported | 22 | 5 | 27
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 8 | 2 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 8 | 9
  White | 27 | 67 | 94
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 3 | 3
Region of Enrollment [Number; unit: participants]
  United States | 36 | 80 | 116

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Overall Survival (OS) at 3 Years
Description: OS defined as the length of time measured from the start of treatment until 3 years post-treatment or death, whichever come first.
Time Frame: 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Surgery (S) vs. SBRT | Stereotactic Body Radiation Therapy (SBRT) (R)
Number analyzed (Participants) | 36 | 80
Participants | 31 | 70

ADVERSE EVENTS:
Time Frame: Adverse Events were assessed after protocol treatment was initiated until three years post-treatment or death, whichever came first.
Arm/Group | Surgery (S) vs. SBRT | Stereotactic Body Radiation Therapy (SBRT) (R)
All-Cause Mortality (participants affected / at risk) | 5/36 | 10/80
Serious Adverse Events (participants affected / at risk) | 3/36 | 8/80
Other Adverse Events (participants affected / at risk) | 3/36 | 3/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Surgery (S) vs. SBRT (N=36) | Stereotactic Body Radiation Therapy (SBRT) (R) (N=80)
Disease progression NOS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 8 (10)
Cardiac ischemia/infarction (Cardiac disorders) | 0 (0) | 1 (1)
Infection-lung (Infections and infestations) | 0 (0) | 1 (1)
Death, NOS (unknown) (Investigations) | 3 (3) | 0 (0)
Infection-Other (sepsis) (Infections and infestations) | 1 (1) | 0 (0)
Infection-Other (COPD/pulmonary) (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Surgery (S) vs. SBRT (N=36) | Stereotactic Body Radiation Therapy (SBRT) (R) (N=80)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Lung fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rib fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-28): https://cdn.clinicaltrials.gov/large-docs/92/NCT02357992/Prot_SAP_000.pdf